CLINICAL TRIAL: NCT04664764
Title: The Effect of Long- and Intermediate-acting Insulins on Glycemic Control and Risk of Hypoglycemia Among Toddlers and Preschool Children With Newly Onset Type 1 Diabetes Mellitus: A Randomized Three Armed Trial
Brief Title: Intermediate and Long Acting Insulin Young Children Type 1 Diabetes.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nouran yousef, Dr, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Basal insulin toddlers
Record Dates: First submitted 2020-12-01; First posted 2020-12-11 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Type 1 Diabetes Mellitus With Hypoglycemia; type1diabetes
MeSH Terms: interventions — insulin degludec; Insulin Glargine; Insulin, Isophane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- degludec arm (Active Comparator): Group A received insulin degludec,
  Interventions: Drug: Degludec
- glargine arm (Active Comparator): group B received insulin glargine
  Interventions: Drug: Glargine
- NPH group (Active Comparator): Group C received NPH insulin
  Interventions: Drug: NPH insulin

INTERVENTIONS:
Drug: Degludec — Basal insulin comparison
  Arms: degludec arm
Drug: Glargine — Basal insulin comparison
  Arms: glargine arm
Drug: NPH insulin — Basal insulin comparison
  Arms: NPH group

SUMMARY:
Background: Achieving glycemic control without risking hypoglycemia imposes a major challenge in the management of toddlers and preschool children with Type 1 diabetes(T1D). Optimal insulin therapy for young children with T1D should provide effective glycemic control while minimizing the risk of hypoglycemia and hyperglycemia. Despite the advantages of the basal-bolus insulin regimens, hypoglycemia still presents a major barrier in achieving desirable glycemic control. Objectives: To compare the effectiveness of insulin degludec to insulin glargine and NPH in toddlers and preschool children with T1D in terms of glycosylated hemoglobin(HbA1C) and frequency of hypoglycemic episodes.

ELIGIBILITY:
Inclusion Criteria:

* Toddlers and preschool children with T1D on insulin therapy

Exclusion Criteria:

* patients with other medical conditions (i.e. celiac disease or autoimmune thyroiditis), patients with other types of diabetes mellitus (i.e. maturity onset diabetes of youth (MODY) and type 2 diabetes mellitus), patients with history of liver disease or any disorder likely to impair liver functions or elevated liver enzymes, renal impairment due to cause other than diabetes, hypertension, patients taking any vitamins or food supplements one month before study and participation in a previous investigational drug study within 3 months preceding screening.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2019-02-21 (Actual); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-03-10 (Estimated)

PRIMARY OUTCOMES:
to compare the effectiveness of insulin degludec to insulin glargine and NPH | 6 months
  to compare the effectiveness of insulin degludec in the form of HBA1C and frequency of hypoglycemia to insulin glargine and NPH in toddlers and preschool children with T1D in terms of HbA1C, IDD and frequency of hypoglycemic episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Safinaz El Habashy, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Data will be available upon request